CLINICAL TRIAL: NCT06121362
Title: Effect of Protocatechuic Acid on Biochemical Markers of Immunity Status in Healthy Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor decided not to pursue
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Raghu Sinha, Associate Professor of Biochemistry and Molecular Biology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STUDY00022594
Record Dates: First submitted 2023-10-29; First posted 2023-11-07 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Immunity
Keywords: dietary supplement, protocatechuic acid, immunity markers
MeSH Terms: interventions — protocatechuic acid; Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Intervention Model Description: We will assign subjects to the placebo or PCA supplementation randomly using Statistical Analysis System (SAS) software that contains a random assignment generator. It will output 50 assignments, equal to the number of subjects that we expect to enroll. Subjects will be assigned to one of the groups in a prospective manner as they are recruited throughout the study period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is a double-blind design. Neither the subject nor the research team will know which treatment arm (placebo or PCA) the enrolled subjects have been assigned to. Study drug bottles will be labeled with a code, and the linked treatment assignment (placebo vs PCA) will be kept with the Sponsor and not made available to the research team during the treatment period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo pill is made of inactive cellulose. Participants will be asked to take 2 capsules daily by mouth in the morning 30 minutes before eating for a total of 14 days (Day 1 - Day 14).
  Interventions: Dietary Supplement: Placebo
- Protocatechuic Acid or PCA (Experimental): Participants will be asked to take 2 capsules (500 mg each of protocatechuic acid or PCA) daily by mouth in the morning 30 minutes before eating for a total of 14 days (Day 1 - Day 14).
  Interventions: Dietary Supplement: Protocatechuic Acid or PCA

INTERVENTIONS:
Dietary Supplement: Protocatechuic Acid or PCA — PCA 1000 mg capsule
  Arms: Protocatechuic Acid or PCA
Dietary Supplement: Placebo — Placebo capsule
  Arms: Placebo

SUMMARY:
The purpose of this voluntary research study is to determine if a dietary supplement containing a substance called protocatechuic acid (PCA) can change markers in blood related to immunity (a body's natural ability to fight diseases and infections) over a 14-day study period. Blood tests and other assessments will be completed before and after taking either 1,000 milligrams a day of protocatechuic acid (PCA) or a placebo (i.e., a sugar pill) for 14 days.

DETAILED DESCRIPTION:
In this pilot study, the Investigator will utilize a double-blind placebo-controlled randomized design. Fifty (50) healthy men and women will be randomized into one of two arms: either agreeing to take placebo or 1000 mg PCA oral capsules daily. Study treatment will continue for 2 weeks (14 days).

At baseline and end of 2 weeks treatment period, various clinical and laboratory measurements will be performed. Vital signs, a 2-chair test, and personal health assessment will be measured, and blood will be drawn. The following endpoints will be evaluated in blood: erythrocyte sedimentation rate (ESR), high sensitivity C-reactive protein (hsCRP), C-X-C motif chemokine ligand 9 (CXCL9), 25-hydroxy vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (i.e., no acute/new symptoms of illness) male and female volunteers
* Ability to provide informed consent and attend study visits
* Adults 50 - 65 years old
* Has not taken any of the following medications in prior 3 months and has no plan to take over the 2-week study period: corticosteroids, anticoagulants (such as aspirin, clopidogrel, heparin, and warfarin), antibiotics, or daily NSAIDs (occasional use is acceptable)
* Has no ill person currently living in household
* Current non-smoker (and has not smoked cigarettes/cigars/pipes or vaped e-cigarettes within the last 6 months)
* Ambulatory without any type of assistance

Exclusion Criteria:

* Cannot provide written informed consent
* Requires assistance ambulating
* Has had any surgery within last 3 months
* Self-report of close exposure to or infection with COVID-19 (with or without symptoms) within last 3 months
* Self-reported history or current status of cancer, uncontrolled diabetes (A1c > 7% or fasting blood glucose of > 140 mg/dL), or heart disease (such as coronary artery disease, arrhythmia, and heart failure)

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Erythrocyte Sedimentation Rate | Baseline and end of 2 weeks
  ESR (mm/hr)
high sensitivity C-Reactive Protein | Baseline and end of 2 weeks
  hsCRP (mg/L)
Chemokine (C-X-C motif) ligand 9 | Baseline and end of 2 weeks
  CXCL9 (ng/mL)
25-hydroxy vitamin D | Baseline and end of 2 weeks
  25-hydroxy vitamin D (ng/mL)

SECONDARY OUTCOMES:
2-Chair test | Baseline and end of 2 weeks
  participant moves 5 times between two chairs placed 5 feet apart, and heart rate and saturation of oxygen (SpO2 %) levels are measured

CONTACTS AND LOCATIONS:
Overall Officials: Raghu Sinha, PhD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No